CLINICAL TRIAL: NCT01406652
Title: One-stage Versus Two-stage Surgical Treatment of Infectious Bursitis
Brief Title: Optimisation of the Treatment of Infectious Bursitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Ilker Uckay, PD Dr. med, MD, Attending, University Hospital, Geneva
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 11-016 (NAC 11-004)
Record Dates: First submitted 2011-06-27; First posted 2011-08-01 (Estimated); Results first posted 2019-11-05 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Olecranon Bursitis; Patellar Bursitis
Keywords: septic bursitis; bursectomy; primary closure

STUDY DESIGN:
Intervention Model Description: Randomization 1:1 with two arms: One versus two-stage bursectomy.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- One-stage bursectomy (Active Comparator): Bursectomy with debridement and primary closure of the wound during one surgical intervention
  Interventions: Procedure: Two-stage bursectomy
- Two-stage bursectomy (Experimental): Bursectomy with debridement and left open. Wound closure in a second step and in a second surgery.
  Interventions: Procedure: Two-stage bursectomy

INTERVENTIONS:
Procedure: Two-stage bursectomy — Debridement, drainage, and secondary closure of septic bursitis during two surgical interventions
  Other Names: There are no "other names"

SUMMARY:
The study investigates prospectively the cost-savings related to a one-stage bursectomy (debridement, drainage and closure at the same time) versus two-stage bursectomy (debridement, left open and closure at a second time) of severe bursitis among hospitalized patients for surgical treatment of septic bursitis.

We suppose that the one-stage bursectomy reveals similar recurrence rates but is associated with a significant shortening of hospital stay, consumption of resources and increased patient satisfaction.

DETAILED DESCRIPTION:
Start as single center interventional study at Geneva University Hospitals Study open for additional centres (electronic CRF) Funding on 24.6.2011 (50,000 Swiss Francs). Further demand for funding ongoing.

Septic bursitis of knee and elbows, for which the patients are hospitalised (a substantial part of patient with failure of conservative treatment) Randomisation 1:1 (one-stage vs. two-stage).

Duration of concomitant postsurgical antibiotic therapy fixed to 7 days Exclusion of severely immuno-depressed patients.

Assessment of all costs of inpatient treatment and outpatient follow-up of included cases.

Interim analysis after ca. 100 cases planified.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Hospitalized for bursectomy for septic bursitis

Exclusion Criteria:

1. Bacteraemic diseases
2. Presence of another concomitant infection requiring antibiotics
3. Presence of osteosynthesis material beneath the bursitis
4. Septic bursitis outside of the elbow or the knee
5. Severe immune suppression (transplantation, HIV with Cluster of Differentiation cell count <200 cells/mm3, immune suppressive treatment with equivalence of more than 15 mg of prednisone daily ).
6. Recurrent septic bursitis episodes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2011-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilker UCKAY, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perez C, Huttner A, Assal M, Bernard L, Lew D, Hoffmeyer P, Uckay I. Infectious olecranon and patellar bursitis: short-course adjuvant antibiotic therapy is not a risk factor for recurrence in adult hospitalized patients. J Antimicrob Chemother. 2010 May;65(5):1008-14. doi: 10.1093/jac/dkq043. Epub 2010 Mar 1. PMID 20197288
- [Background] Uckay I, von Dach E, Perez C, Agostinho A, Garnerin P, Lipsky BA, Hoffmeyer P, Pittet D. One- vs 2-Stage Bursectomy for Septic Olecranon and Prepatellar Bursitis: A Prospective Randomized Trial. Mayo Clin Proc. 2017 Jul;92(7):1061-1069. doi: 10.1016/j.mayocp.2017.03.011. Epub 2017 Jun 8. PMID 28602435
- [Background] Baumbach SF, Wyen H, Perez C, Kanz KG, Uckay I. Evaluation of current treatment regimens for prepatellar and olecranon bursitis in Switzerland. Eur J Trauma Emerg Surg. 2013 Feb;39(1):65-72. doi: 10.1007/s00068-012-0236-4. Epub 2012 Nov 8. PMID 26814924

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: See below
Groups:
- One-stage Bursectomy: 79 patients undergo surgical bursectomy and wound closure within the same Operation.
- Two-stage Bursectomy: 85 patients have a two-stage Approach. First, they undergo surgical bursectomy with the wound left open. In a second step 3-4 days later, they are re-operated for wound closure.
Period: Overall Study
Arm/Group | One-stage Bursectomy | Two-stage Bursectomy
Started | 109 | 115
Completed | 89 | 95
Not Completed | 20 | 20
Not completed — Lost-to-follow-up | 3 | 4
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Insufficient follow-up | 5 | 4
Not completed — Infection not sure | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | One-stage Bursectomy | Two-stage Bursectomy | Total
Number analyzed (Participants) | 79 | 85 | 164
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 80 | 150
  >=65 years | 9 | 5 | 14
Age, Continuous [Median (Full Range); unit: years] | 53 [18 to 94] | 51 [20 to 86] | 52 [18 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 11 | 28
  Male | 62 | 74 | 136
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 79 | 85 | 164
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Switzerland | 79 | 85 | 164

OUTCOME MEASURES:

1. Primary Outcome: Overall Costs of the Combined Surgical and Medical Treatment
Description: The overall costs are of primary interest in the study protocol.
Time Frame: 2 months
Population: The overall costs (Swiss francs; CHF) are of primary interest in the study protocol
Measure: Median (Inter-Quartile Range); unit: Swiss Francs
Groups:
- One-stage Bursectomy; Two-stage Bursectomy: Total costs in Swiss francs of the one-stage bursectomy approach and associated treatment.
Arm/Group | One-stage Bursectomy | Two-stage Bursectomy
Number analyzed (Participants) | 79 | 85
Swiss Francs | 6881 [4587 to 8254] | 11178 [9231 to 12498]

2. Secondary Outcome: Number of Participants With Post-surgical Wound Dehiscence
Description: We assess clinical failures of bursectomy for bursitis. As recurrences are associated with wound dehiscence, we evaluate the dehiscence a the most important parameter for Failure. Of course, dehiscence can also occur without recurrent infection, but this is also considered as failure.
Time Frame: 2 months
Measure: Number; unit: participants
Arm/Group | One-stage Bursectomy | Two-stage Bursectomy
Number analyzed (Participants) | 79 | 85
participants | 2 | 10

ADVERSE EVENTS:
Time Frame: 2 months post surgical follow-up
Groups:
- One-versus Bursectomy: Bursectomy and surgical wound closure during the same surgery
- Two-stage Busectomy: Bursectomy during the first surgery, followed by a surgical closure in a second step.
Arm/Group | One-versus Bursectomy | Two-stage Busectomy
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/85
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/85
Other Adverse Events (participants affected / at risk) | 14/79 | 15/85
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | One-versus Bursectomy (N=79) | Two-stage Busectomy (N=85)
Handicap (Musculoskeletal and connective tissue disorders) | 14 (14) | 15 (15) — Persistant postsurgical pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes